CLINICAL TRIAL: NCT06600074
Title: Effect of Retro-walking on Postpartum Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safa Magdy Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004491
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Disorder; Low Back Pain
MeSH Terms: conditions — Puerperal Disorders; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back care advice + Postural correction exercises (Active Comparator): It will include 18 postpartum women who will receive back care advice and postural correction exercises.
  Interventions: Behavioral: Back care advice; Other: Postural correction exercises
- Back care advice + Postural correction exercises + Retro-walking (Experimental): It will include 18 postpartum women who will receive the same back care advice and postural correction exercises, in addition to retro-walking.
  Interventions: Behavioral: Back care advice; Other: Postural correction exercises; Other: Retro-walking

INTERVENTIONS:
Behavioral: Back care advice — All patients in both groups will be advised to use proper lifting techniques, avoid prolonged sitting or standing, maintain a healthy weight, quit smoking, practice good posture, take breaks, spread housekeeping duties over the whole week, and sleep in supportive positions.
Other: Postural correction exercises — All patients in both groups will be instructed to perform postural correction exercise. They will be performed from different positions (crock lying, supine lying, supine, sitting and standing position). They will lie in crock lying position for example and the physical therapist will instruct them to do chin in , open out ribs through costal breathing, contract abdominal muscles, contract glutei, hold for 6 seconds and relax and repeat 10 times.
Other: Retro-walking — Patients in the experimental group only will practice walking backward on a treadmill, starting with a 5-minute warm-up at a self-selected speed, then gradually increasing speed from 1.2 to 1.6 m/s based on comfort and progress.
  Arms: Back care advice + Postural correction exercises + Retro-walking

SUMMARY:
This study will be conducted to determine the effect of retro walking on post partum low back pain.

DETAILED DESCRIPTION:
Postpartum LBP is a common musculoskeletal disorder. It occurs due to ligament laxity and postural changes that started during pregnancy or within 3 weeks of childbirth and continue for 3 months after delivery. When all forms of non-specific LBP were considered, approximately 33% of postpartum women had some LBP within 3 months after childbirth, and approximately 40% described moderate to severe disability.

Postpartum LBP stresses the sacroiliac joints and lumbosacral spine. Previous studies of Swedish women with postpartum LBP reported impairments to their daily activities with a prevalence ranging between 20-90%, but they seldom sought health care assistance or treatment.

Many researchers and clinicians have suggested that an increase in core strength and improvement in pelvic alignment are keys to resolve or avoid LBP. During backward walking, the typical heel-strike associated with ground contact is eliminated because the toe contacts the ground first and the pelvis is anteriorly aligned. This may open up the facet joints in the vertebral column and help in alleviating the pressure on intervertebral discs and the associated LBP.

Previous studies investigated the effect of retro walking on other types of LBP (non-specific and chronic) but till now, there is no previous study investigate the effect of retro walking on postpartum LBP related to C.S delivery. So, this study will be the first one in this issue. Therefore, this study will be of valuable benefits for medical service organization and increase the body of knowledge in physical therapy field.

ELIGIBILITY:
Inclusion Criteria:

* Multi parous women suffering from postpartum low back pain after cesarean delivery (from 6 weeks to 6 months after delivery).
* Their ages will range from 25-35 years old.
* Their body mass index will be less than 30 Kg/m2.
* They should have mild to moderate low back pain as scored on VAS (represented by cut points on the scale recommending mild pain (5- 44mm), moderate pain (45- 74mm))

Exclusion Criteria:

* Recent surgeries, trauma or fractures of the lower limb or in the back region.
* Morbid cardiovascular disease.
* Liver or kidney dysfunction.
* Any neurological disorders including balance issues or motor and sensory loss.
* Any musculoskeletal disorders such as disc prolapsed, lumbar canal stenosis and spondylysthesis or severe knee osteoarthritis.
* Taking intra-articular injection for knee for the last 6 months.
* Those having visual dysfunction or refractory errors not corrected with glasses or contact lenses.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 6 weeks
  It will be used to measure the severity of post cesarean low back pain before and after the treatment program for all participants in both groups. The VAS is ten cm horizontal line on which the patients' pain intensity is represented by a point between the extremes of no pain at all (no pain=0) and worst pain imaginable (worst pain=10). Each participating woman will be asked to put a mark on the line at the point indicating her pain level / intensity.
Lumbar flexion range of motion (ROM) | 6 weeks
  It will be assessed by the Modified Schober test before and after the treatment program for all participants in both groups. The therapist will mark the lumbar spine at the posterior superior iliac spines, with another mark 15 cm above it. A tape measure will be used to record the distance between the marks in a standing position, then again after the patient bends forward into full lumbar flexion. The difference indicates the lumbar flexion ROM. This test will be repeated three times, and the average value will be taken as the lumbar flexion ROM.
Lumbar extension range of motion (ROM) | 6 weeks
  It will be assessed by the Modified Schober test before and after the treatment program for all participants in both groups. The therapist will mark the lumbar spine at the posterior superior iliac spines, then place another mark 15 cm above. A tape measure will record the distance between the marks while the patient is standing. The patient will then bend backward into full lumbar extension, and the new distance between the marks will be measured. The difference represents the lumbar extension ROM. This process will be repeated three times, with the average value taken as the lumbar extension ROM.

SECONDARY OUTCOMES:
Oswestry disability questionnaire | 6 weeks
  It will be used to assess functional disability for all women in both groups before and after the end of the treatment program. The Oswestry disability questionnaire is considered the "gold standard" tool for low back functional outcome It is consisted of 50 questions covering 10 sections (personal care, lifting, sitting, standing, walking, sex life, sleeping, social life and travelling). Each question is scored from 0-5, giving maximum score of 50 if one section is missed, the total score will be 45 and then the score is converted into percentage. scores are classified according to severity into minimal disability (10-20%), moderate disability (21-40%), sever disability (41-60%) crippled (61-80%) and bed bound (81-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Mohamed Mahmoud Botla, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Giza, Egypt